CLINICAL TRIAL: NCT00960726
Title: Phase 2 Study of NOV-002 in Low and Intermediate-1 Risk Myelodysplastic Syndrome
Brief Title: NOV-002 in Myelodysplastic Syndrome (MDS)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn at sponsor request.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0673
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia; Myelodysplastic Syndrome
Keywords: Leukemia; NOV-002; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — NOV 002

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOV-002 (Experimental)
  Interventions: Drug: NOV-002

INTERVENTIONS:
Drug: NOV-002 — 60 mg delivered daily subcutaneously for up to 12 months.

SUMMARY:
The goal of this clinical research study is to learn if NOV-002 can help to restore bone marrow and blood levels in patients who have MDS. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

NOV-002 is a type of blood cell production stimulating drug. NOV-002 is believed to stimulate the bone marrow to increase production of mature cells in the bloodstream, including red and white blood cells and platelets.

Screening Tests:

Signing this consent form does not mean that you will be able to take part in this study. You will have "screening tests" to help the doctor decide if you are eligible to take part in this study. The following tests and procedures will be performed:

* Your medical history will be recorded.
* You will be asked about any drugs you have taken or may be taking.
* You will have a physical exam, including measurement of your weight and vital signs (blood pressure, temperature, breathing rate, and heart rate).
* Urine will be collected for routine tests.
* Blood (about 7 teaspoons) will be drawn for routine tests and to check for HIV and hepatitis B and C.
* If you have not had a bone marrow aspiration in the month before the screening tests, one will be performed to check the status of the disease. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.
* Women who are able to become pregnant will have a pregnancy test as part of the routine blood or urine collection. To take part in this study, the pregnancy test must be negative.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive the study drug NOV-002 through a needle under the skin 1 time each day while you are on study.

The study staff will teach you and/or a caregiver how to inject the study drug. The study staff will also give you written copy of instructions on how and when you should inject the study drug.

You will be given diary cards to record when and where on your body you inject the study drug, as well as any side effects that may occur. If you miss a dose of study drug, you should note that on your diary card and take the study drug the next day as scheduled. You should not take a double, "make-up" dose at that time.

You must store the study drug in a refrigerator and out of the reach of children. You will be asked to bring all leftover study drug to each study visit.

Study Visits:

* You will have study visits 1 time each week during Weeks 1-8 and 1 time each month during Months 3-12. At these visits, the following tests and procedures will be performed:
* You will be asked about any drugs you have taken or may be taking and about any side effects you may have experienced.
* Your vital signs will be measured.
* Blood (about 5 teaspoons) will be drawn for routine tests.
* You will have a physical exam 1 time each month while you are on study.
* You will have a bone marrow aspiration every 3 months while you are on study to check the status of the disease.

Length of Study:

You will take the study drug for up to 12 months. You will be taken off study if you have intolerable side effects, if the disease gets worse, or if the doctor thinks it is in your best interest.

Long-Term Follow-Up:

After you have finished taking the study drug for any reason, the following procedures will be performed for about 12 months, but will be stopped if you start receiving a different treatment or if the disease gets worse:

Blood (about 5 teaspoons) will be drawn for routine tests 1 time each month. You will have a bone marrow aspiration every 3 months.

This is an investigational study. NOV-002 is not FDA approved or commercially available. At this time, it is only being used in research.

Up to 40 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years
2. Women of child-bearing potential and men whose partners are of child-bearing potential must be willing to use an acceptable method of birth control during trial participation or are surgically sterile or women who are post-menopausal (defined as not having a menstrual cycle for greater than two years). Acceptable methods of birth control are: cervical cap or diaphragm with spermicide, condom, oral birth control pills, intrauterine device (IUD), or implanted or injectable birth control.
3. The patient must have the ability to understand and the willingness to sign a written informed consent form and agree to abide by the trial restrictions and to return for the required assessments
4. The patient must be able to self administer daily subcutaneous injections or their caregiver must be able to administer daily subcutaneous injections
5. Has a diagnosis of myelodysplastic syndrome and IPSS score of less than or equal to 1
6. Documented cytopenias persistent for 2 months defined as:

   * Red cell transfusion dependence defined as receiving 4 or more units of red cells within a period of 8 weeks for anemia of hemoglobin less than 9 gm/dL; and/or
   * Untransfused hemoglobin of 10 gm/dL or less on two occasions greater than or equal to 1 week apart; and/or
   * Platelet count less than 50 x 10(9) /dL on two occasions greater than or equal to 1 week apart; and/or
   * Neutropenia defined as ANC less than 1 x 10(6) /dL on two occasions greater than or equal to 1 week apart.
7. Adequate organ function defined as:

   * Bilirubin less than or equal to 2.5 mg/dL (unless clearly attributable to hemolysis);
   * Creatinine less than or equal to 2mg/dL or calculated creatinine clearance greater than 50 ml/min;
   * AST or ALT less than 3 times the upper limit of institutional normal (ULN).
8. Must have discontinued any growth factor for a period of 3 weeks prior to enrollment
9. Up to one prior conventional or experimental therapy for MDS (not including growth factors and transfusion) is allowed but there must be a washout of 4 weeks prior to enrollment from any such therapy (examples include lenalidomide, hypomethylating agent etc.)

Exclusion Criteria:

1. Pregnant female or nursing mother
2. Active second malignancy excluding carcinoma in-situ of uterine cervix, basal or squamous cancer of skin
3. Active hepatitis B or C infection
4. Known HIV positive
5. On oral steroids (prednisone or equivalent) greater than 10 mg/day
6. NOV-002 is contraindicated in patients with known hypersensitivity to any of the components of NOV-002

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Overall Response (OR) | Baseline to measured progressive disease (anticipated treatment period 3 -12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MBBS, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org